CLINICAL TRIAL: NCT02567201
Title: Electrophysiological Evaluation of Voluntary Attention
Acronym: EVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL15_0216; 2015-A00635-44 (Other: ID-RCB)
Record Dates: First submitted 2015-09-28; First posted 2015-10-02 (Estimated); Last update posted 2024-12-24 (Actual); Status verified 2024-02

CONDITIONS: Brain Injury
Keywords: Voluntary attention; Electroencephalogram; Brain-computer interface; Disorders of consciousness
MeSH Terms: conditions — Brain Injuries; Consciousness Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Electrophysiological assessment of Healthy subjects (Experimental): Experiences 1, 2 and 3 with healthy subjects
  Interventions: Other: electrophysiological evaluation
- Electrophysiological assessment of patients (Experimental): Experiences 1, 2 and 3 with patients
  Interventions: Other: electrophysiological evaluation of patients

INTERVENTIONS:
Other: electrophysiological evaluation — electrophysiological assessment (experience 1 : passive ; experience 2 : active versus passive ; experience 3 : active, with feedback) Experience 1, 2, 3 : one session maximum by experience
  Arms: Electrophysiological assessment of Healthy subjects
Other: electrophysiological evaluation of patients — electrophysiological assessment (experience 1 : passive ; experience 2 : active versus passive ; experience 3 : active, with feedback) Experience 1 : maximum one session by sensory modality of stimulation (auditory, tactile, or visual) Experience 2 : maximum one session by sensory modality of stimulation (auditory, tactile, or visual) Experience 3 : Stimulation = auditory or visual ; possibility of several sessions if the patient is tired.
  Arms: Electrophysiological assessment of patients

SUMMARY:
Aim : To assess the ability of healthy subjects and patients with a severe motor disability to voluntary control their attention

Material and Methods:

Population: healthy subjects, patients with brain injury Electroencephalographic study to research attentional modulation during different kind of stimulation (visual, auditory, tactile)

Sudy 1: passive recording.

Study 2: active recording (instruction of attentional control given to the subject).

Study 3: active recording with a feedback obtained after a processing of the brain activity.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for patients :

* Adults, man or woman, left or right-handed, from 18 years old to 80 years-old ;
* Diagnosis :

  * Locked-in syndrome :

< Brainstem injury, without any evolution for at least 3 week, etiology : vascular, traumatic < Amyotrophic Lateral Sclerosis < Following damage to the central or peripheral nervous system

* Or Minimal conscious state or Unresponsive Wakefulness Syndrome consecutive to a severe acquired brain injury for at least one month
* Or with a severe brain injury, since birth or acquired, for at least one month
* Or with Guillain-Barré syndrome

  * Subjects affiliated to social security;
  * Signature of consent form by the patient or by a relative (family member or "the trusted person") if obtaining a consent is impossible

Inclusion criteria of Healthy subjects

* Adults, man or woman, left or right-handed, from 18 years old to 80 years-old ;
* Without known auditory impairment
* Subjects able to understand the experimental instructions
* Subjects affiliated to social security;
* Signature of consent form

Exclusion criteria of patients and healthy subjects

* Medical history : psychiatric disorders (except if due to brain injury), neurologic disorders (except if due to brain injury)
* For healthy subjects : history of brain injury
* Pregnant women or breastfeeding women
* Person under legal protection
* Medico-legal conflicts
* Absence of consent by the subject or the patient or his/her representant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2015-10-16 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
Research of statistical differences between sensory evoked potentials in attentional oriented condition and distracted condition | through study completion, an average of 3 years
  stastical analysis allowing to compare evoked responses during different stimulation condition (attentionnaly oriented versus attentionnally distracted versus passive condition = no instruction to the subject). These comparisons are made either for one single subject and at the group level. Analysis mainly concerns the differences in amplitude variation between the differents evoked potentials on several electrods of interest. These can vary between patients because of the different topographies of lesions and because of the different adaptative strategies. The statiscal difference will be assessed by a randomization test (also called "permutation test") wich allow to assess how high is the risk that the observed difference between the evoked potential (amplitude, variance) is due to chance or not

SECONDARY OUTCOMES:
Online and offline accuracy | through study completion, an average of 3 years.
  percentage of correct answers with the brain-computer interface (BCI). A "correct answer" is recorded each time the feedback of the BCI match the command sended by the subject controlling the BCI. This analysis can be done online and offline. Online accuracy is recorded in real-time during the session with the subject. offline accuracy is obtained a posteriori of the experiment, to test the impact on accuracy of the changes in different parameters (stimuli duration, numbers of spatial filtering, change of classifiers, etc.).
Clinical scale score ("Evaluation de la Communication des patients en Eveil de Coma" (ECEC) scale) | an average of 3 years (At the group level)
  this clinical scale allow to obtain an outcome measure of the investissment, the communication themes and the communication modes of the patient. The final global value range between 0 and 44.

CONTACTS AND LOCATIONS:
Overall Officials: Jacques LUAUTE, MD, Principal Investigator — Hospices Civils de Lyon
Locations (11):
- France (11):
  - Centre Médical de L'argentière, Aveize
  - Centre Hospitalier Georges Claudinon, Le Chambon-Feugerolles
  - Hospices Civils de Lyon, Lyon
  - Centre de Recherche en Neurosciences de Lyon, Lyon
  - CHU de Nantes, Nantes
  - CHU de Nîmes, Nîmes
  - APHP - Hôpital de la Pitié Salpêtrière, Paris
  - APHP - Hôpital Raymond Poincaré, Paris
  - Hôpital Nord CHU Saint Etienne, Saint-Etienne
  - Hospices civils de Lyon, Hôpital Henry Gabrielle,, Saint-Genis-Laval
  - Centre Médical Germaine Revel, Saint-Maurice-sur-Dargoire

REFERENCES:
- [Derived] Seguin P, Maby E, Fouillen M, Otman A, Luaute J, Giraux P, Morlet D, Mattout J. The challenge of controlling an auditory BCI in the case of severe motor disability. J Neuroeng Rehabil. 2024 Jan 18;21(1):9. doi: 10.1186/s12984-023-01289-3. PMID 38238759